CLINICAL TRIAL: NCT02558556
Title: Near-infrared Fluorescence Cholangiography Assisted Laparoscopic Cholecystectomy Versus Conventional Laparoscopic Cholecystectomy (FALCON): a Multicenter Randomized Controlled Trial
Brief Title: FALCON: a Multicenter Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL47718.068.14
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Cholecystolithiasis; Cholecystitis
Keywords: Laparoscopic cholecystectomy (LC); Indocyanine green (ICG); Near-Infrared Fluorescence Imaging (NIRF); Critical View of Safety (CVS)
MeSH Terms: conditions — Cholecystolithiasis; Cholecystitis | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIRF-LC (Experimental): This group of patients will undergo near-infrared fluorescence cholangiography assisted laparoscopic cholecystectomy by use of a Laparoscopic Fluorescence Imaging System (Karl Storz), in combination with one intravenous injection of contrast agent ICG. The ICG is given directly after induction of anesthesia in a dose of 1 ml of 2,5 mg/ml solution.
  Intraoperatively every 2-5 minutes (more often if desired by surgeon) camera is switched to ICG mode for fluorescence cholangiography, until CVS is established.
  Registration of time until establishment of CVS, visualization of the individual structures as described as secondary endpoints, and total operation time will be done.
  The complete procedure will be recorded on video.
  Interventions: Device: Laparoscopic Fluorescence Imaging System (Karl Storz); Other: Indocyanine Green
- CLC (No Intervention): This group will undergo conventional laparoscopic cholecystectomy as in standard practice with no other intervention.
  Registration of time until establishment of CVS, visualization of the individual structures as described as secondary endpoints, and total operation time will be done.
  The complete procedure will be recorded on video.
  Postoperatively, as in the NIRF-LC arm, the videos will be analysed to determine whether CVS is actually established, is the transition of the cystic duct into the gallbladder visualized? Is transition of the cystic artery into the gallbladder visualized? Furthermore, cost-minimalisation will be calculated.

INTERVENTIONS:
Device: Laparoscopic Fluorescence Imaging System (Karl Storz) — The Laparoscopic Fluorescence Imaging System (incl. laparoscope, light source, light cable) will supply the needs for near-infrared fluorescence imaging with ICG. The hypothesis is that this device will help in visualizing the anatomical structures such as the common bile duct, which are hard to visualize in white light due to the surrounding tissues.
  Arms: NIRF-LC
Other: Indocyanine Green — Indocyanine Green will be injected intravenously as a contrast agent for the use of the Laparoscopic Fluorescence Imaging System.
  Other Names: ICG
  Arms: NIRF-LC

SUMMARY:
Rationale: Several clinical feasibility studies have shown the potential benefit of near-infrared fluorescence (NIRF) imaging using indocyanine green (ICG) for enhanced and earlier biliary anatomy visualization during laparoscopic cholecystectomy with the aim to reduce the number of vascular and biliary injuries. Although the incidence of injuries is low (0.7%), the impact on patients in terms of morbidity, quality of life and costs are dramatic. The Critical View of Safety (CVS) technique is regarded as the safety valve in conventional laparoscopic cholecystectomy (CLC). It is hypothesized that standard application of near-infrared fluorescence imaging during laparoscopic cholecystectomy can be useful to obtain establishment of CVS (at least 5 minutes) earlier and with more certainty regarding visualization when compared to conventional laparoscopic imaging alone.

Study design: A multicenter randomized controlled trial with two study arms. Patients scheduled for an elective laparoscopic cholecystectomy will be recruited and randomized at the outpatient clinic (n = 308 total). One group will undergo near-infrared fluorescence cholangiography assisted laparoscopic cholecystectomy (NIRF-LC) and the other group will undergo conventional laparoscopic cholecystectomy (CLC).

Compared with standard care, patients in the NIRF-LC group have to receive one preoperative intravenous injection of ICG. This is the only additional minimally invasive action for the patient. Initially, patients participating in this study will not benefit from the application of NIRFC during the surgical procedure. The administration of ICG and the modified laparoscope itself are not related with any kind of additional risk for the patient.

Despite the encouraging results from several (pre)clinical feasibility studies, wide clinical acceptance of the routine use of ICG fluorescence laparoscopy is still lacking due to the absence of reliable and validated clinical data. A randomized clinical study is desirable to assess the potential added value of the NIRF imaging technique during laparoscopic cholecystectomy. Strong evidence in favor of routine implementation of this new imaging technique during laparoscopic cholecystectomy, will probably lead to worldwide routine application of the NIRF technique. Therewith long term sustainability of this research project is guaranteed.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is one of the most commonly performed laparoscopic procedures in gastrointestinal surgery. Bile duct injury during this procedure is rare but constitutes a serious complication (0.3-0.7%) (Flum 2003, Fletcher 1999, Nuzzo 2005 and Waage 2005). Misidentification of the extra-hepatic bile duct anatomy during laparoscopic cholecystectomy is the main cause of bile duct injury (Way 2006).

The Critical View of Safety (CVS) technique, which was first described by Strasberg in 1995 (Strasberg 2003) and recommended by the Dutch Guidelines and Best Practice for laparoscopic cholecystectomy (Lange 2006), was introduced to reduce the risk of bile duct injury. To establish CVS, two windows need to be created: one window between the cystic artery, cystic duct and gallbladder, another window between the cystic artery, gallbladder and liver. The CVS technique is especially aimed at mobilizing the gallbladder neck from the liver, in order to obtain a circumferential identification of the transition of the cystic duct into the gallbladder.

Intraoperative cholangiography has been advised to reduce the risk of bile duct injury (Flum 2003, Buddinhg 2011). However, this radiological imaging of the biliary tree is only used selectively, as the process takes time, radiation exposure is involved and additional equipment and manpower for the procedure are required. Therefore, worldwide consensus about implementation of intraoperative cholangiography is still lacking (Ford 2012).

Near-infrared fluorescence (NIRF) imaging after intravenous injection of indocyanine green (ICG) is a promising new technique for easier intraoperative recognition of the biliary anatomy. It may help improve the outcome of laparoscopic cholecystectomy (Buddingh 2011, Agarwal 2009). ICG is cleared quickly and exclusively by the liver after intravenous administration. Neither radiological support nor additional intervention, such as opening the biliary tree, is required. The NIRF laparoscopy technique using ICG has been evaluated in various animal models (Figueiredo 2010, Figueiredo 2011, Tagaya 2010, Matsui 2010) and in open, laparoscopic, and single-incision laparoscopic cholecystectomy (Tagaya 2010, Ishazawa 2010, Ishazawa 2011 Aoki 2010). Promising results were presented for successful intraoperative identification of the common bile duct and the cystic duct, compared to conventional laparoscopic imaging. Another clinical study showed that the NIRFC technique provides significantly earlier identification of the extra-hepatic bile ducts during the CVS dissection phase: up to 10 minutes earlier identification of cystic duct and common bile duct could be obtained (Schols 2012). Real-time simultaneous imaging of the hepatic and cystic arteries can also be obtained (Ashitate 2011, Mitsuhashi 2008, Schols 2013).

Despite the encouraging results from these (pre)clinical feasibility studies, wide clinical acceptance of the routine use of ICG fluorescence laparoscopy is still lacking due to the absence of reliable clinical data. Therefore, a multicenter randomized clinical study is desirable to assess the potential added value of the fluorescence imaging technique during laparoscopic cholecystectomy in order to perform a more safe procedure leading to a reduction in the vascular and bile duct injuries. This study will compare NIRF assisted laparoscopic cholecystectomy to conventional laparoscopic cholecystectomy.

The main objective of this study is to evaluate whether earlier establishment of Critical View of Safety can be obtained using the NIRF laparoscopy technique during laparoscopic cholecystectomy. This will shorten the operation time, and thereby reduce the cost of the procedure.

Study design: Multicenter randomized controlled trial. 308 patients will be included for randomization. All patients (age >18 years) scheduled for an elective laparoscopic cholecystectomy and meeting the inclusion criteria will be suitable for inclusion. Patients will be included in at least 3 hospitals in The Netherlands: Maastricht University Medical Center+; Leiden University Medical Center; Catharina Hospital.

Treatment of subjects: All operations will be performed by a surgical resident, assisted by a surgeon or surgical resident with a track record of at least 50 laparoscopic cholecystectomies, or will be performed by a surgeon or surgical resident with that track record him/herself. In the CLC group conventional laparoscopic cholecystectomy will be performed using conventional laparoscopic imaging systems. In the NIRF-LC group, using laparoscopic fluorescence imaging systems near-infrared fluorescence cholangiography technique will be conducted to assist during laparoscopic cholecystectomy. To obtain fluorescence imaging of the biliary tract a contrast agent has to be administered. Directly after induction of anesthesia the fluorescent dye, indocyanine green (ICG), will be administered for intraoperative visualization of the extra-hepatic bile ducts with the NIR fluorescence laparoscope. Since many years ICG has been approved for commercial and clinical diagnostic use by the FDA.

Randomization: After inclusion in the study (i.e., after written informed consent is obtained) patients will be randomized to NIRF-LC or CLC group. Randomization will be performed centrally. Computerized treatment allocation will be conducted on the day of surgery. There will be no blinding of patients or surgeons.Stratification factor will be performed for participating center.The experience level of the surgical team will be recorded, but no stratification will take place for this factor, as due to the large volume of patients an even distribution of skill level over both randomization arms in expected. Experience is defined in performing laparoscopic cholecystectomy as first surgeon.

Study procedures: The laparoscopic cholecystectomy procedure itself will not be performed differently than usual. Next, there will not be any radiation involved for the patient. Neither are any psychological or psychiatric investigations involved. Patients are not asked to undergo additional testing after the surgical procedure, they are also not requested to fulfill any questionnaire.

The following procedures will be conducted during this study:

* Preoperative (NIRF-LC group): Directly after induction of anesthesia 1ml (2,5mg/ml) indocyanine green will be administrated via intravenous injection, by the surgeon or surgical trainee (under supervision of the surgeon and the anesthesiologist).
* Intraoperative (CLC and NIRF-LC group): Intraoperatively the PhD researcher / local researcher (to be appointed in each participating center) systematically whether the localization of the common bile duct, cystic duct and cystic artery can be identified at set time points, by both the conventional camera mode (CLC group) and fluorescence camera mode (NIRF-LC group). Also establishment of CVS is registered. For agreement on the identification of the aforementioned structures the attending surgeon is consulted. A structure is scored as 'identified' if its localization is confirmed with great certainty by the experienced surgeon. In case of the common bile duct this does explicitly not mean that it was surgically exposed, as this is contradictory to the CVS-technique. In accordance with regular care, all laparoscopic surgical procedures will be digitally recorded.
* Postoperative qualitative video analysis (CLC and NIRF-LC group)

Performed by expert panel of 3 surgeons:

* Is CVS actually established? (and: at what time is CVS established?)
* Time until identification of the cystic duct, and time until identification of the transition of the cystic duct in the gallbladder during dissection of CVS;
* Time until identification of the cystic artery, and time until identification of the transition of the cystic artery in the gallbladder during dissection of CVS; Postoperative quantitative fluorescence image analysis (NIRF-LC group): For objective assessment of the degree of fluorescence illumination in the extra-hepatic bile ducts and artery, OsiriX 5.5.1 Imaging Software will be used. The fluorescence images will be analyzed by determining target-to-background ratio (TBR). TBR is defined as the mean fluorescence intensity (FI) of two point regions of interest (ROIs) in the target (i.e. CBD, CD or CA) minus the mean fluorescence intensity of two background (BG) ROIs in the liver hilum, divided by the mean fluorescence intensity of the two background ROIs in the liver hilum; in formula: TBR = (FI of target - FI of BG) / FI of BG.

Postoperative registration of secondary endpoints (CLC and NIRF-LC group). The researcher will document the following remaining secondary endpoints: Intraoperative bile leakage from the gallbladder or cystic duct; Bile duct injury; Postoperative length of hospital stay; Complications due to the intravenously injected contrast agent; Conversion to open cholecystectomy; Postoperative complications (until 90 days after surgery) After 90 days the patient will contacted by telephone to register any complications that occurred after the routine visits.

Cost-effectiveness minimisation of the procedure will be calculated, limited to the per-operative period. The observed reduction in time until CVS, calculated in cost per minute use of the operating suite, will be weighed against the extra cost of the use of the equipment and the fluorescent dye.

Postoperative analysis of time measurements (CLC and NIRF-LC group) Regarding the primary and secondary endpoints, a linear regression analysis will be applied for determination of possible significant differences between the time measurements from "first look at liver hilum" until "establishment of CVS" / "identification of transition CD in gallbladder" / "identification of transition CA in gallbladder"; therewith comparing fluorescence laparoscopic imaging with conventional laparoscopic imaging. In case of missing values (which can occur with the expert panel analysis, when the panel concludes that actually no CVS was obtained or the transition of the mentioned structures in the gallbladder had not been properly identified) a Cox regression analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective laparoscopic cholecystectomy
* Normal liver and renal function
* No hypersensitivity for iodine or ICG
* Able to understand nature of the study procedures
* Willing to participate and with written informed consent
* Physical Status Classification: ASA I / ASA II

Exclusion Criteria:

* Age < 18 years
* Liver or renal insufficiency
* Known iodine or ICG hypersensitivity
* Pregnancy or breastfeeding
* Not able to understand nature of the study procedure
* Physical Status Classification: ASA III and above
* iv Heparin injection in the last 24 h; (LMWH not contraindicated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
time to identification of CVS | at time of surgery
  change in time to identification of CVS

SECONDARY OUTCOMES:
time until identification of the transition of the cystic duct in the gallbladder during dissection of CVS | at time of surgery
  change in time to identification
visualization of CVS and visualization of the transition of the cystic duct and cystic artery in the gallbladder | at time of surgery
  Are these structures actually visualized?
total surgical time | at time of surgery
  change in duration of surgery
intraoperative bile leakage from the gallbladder or cystic duct | at time of surgery
  change in number of intraoperative bile leakage from the gallbladder or cystic duct
bile duct injury | up to 90 days
  change in number of bile duct injuries
postoperative length of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 1-2 days
  change in length of hospital stay
complications due to the injected contrast agent | at time of surgery
  appearance of complications in intervention group
conversion to open cholecystectomy | at time of surgery
  change in number of conversions
postoperative complications | up to 90 days
  change in number of postoperative complications
cost-minimisation: difference in costs between the treatment in both groups | up to 90 days
  change in costs per patient

CONTACTS AND LOCATIONS:
Overall Officials: Laurents PS Stassen, MD, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Flum DR, Dellinger EP, Cheadle A, Chan L, Koepsell T. Intraoperative cholangiography and risk of common bile duct injury during cholecystectomy. JAMA. 2003 Apr 2;289(13):1639-44. doi: 10.1001/jama.289.13.1639. PMID 12672731
- [Background] Fletcher DR, Hobbs MS, Tan P, Valinsky LJ, Hockey RL, Pikora TJ, Knuiman MW, Sheiner HJ, Edis A. Complications of cholecystectomy: risks of the laparoscopic approach and protective effects of operative cholangiography: a population-based study. Ann Surg. 1999 Apr;229(4):449-57. doi: 10.1097/00000658-199904000-00001. PMID 10203075
- [Background] Nuzzo G, Giuliante F, Giovannini I, Ardito F, D'Acapito F, Vellone M, Murazio M, Capelli G. Bile duct injury during laparoscopic cholecystectomy: results of an Italian national survey on 56 591 cholecystectomies. Arch Surg. 2005 Oct;140(10):986-92. doi: 10.1001/archsurg.140.10.986. PMID 16230550
- [Background] Waage A, Nilsson M. Iatrogenic bile duct injury: a population-based study of 152 776 cholecystectomies in the Swedish Inpatient Registry. Arch Surg. 2006 Dec;141(12):1207-13. doi: 10.1001/archsurg.141.12.1207. PMID 17178963
- [Background] Way LW, Stewart L, Gantert W, Liu K, Lee CM, Whang K, Hunter JG. Causes and prevention of laparoscopic bile duct injuries: analysis of 252 cases from a human factors and cognitive psychology perspective. Ann Surg. 2003 Apr;237(4):460-9. doi: 10.1097/01.SLA.0000060680.92690.E9. PMID 12677139
- [Background] Strasberg SM, Hertl M, Soper NJ. An analysis of the problem of biliary injury during laparoscopic cholecystectomy. J Am Coll Surg. 1995 Jan;180(1):101-25. No abstract available. PMID 8000648
- [Background] Buddingh KT, Nieuwenhuijs VB, van Buuren L, Hulscher JB, de Jong JS, van Dam GM. Intraoperative assessment of biliary anatomy for prevention of bile duct injury: a review of current and future patient safety interventions. Surg Endosc. 2011 Aug;25(8):2449-61. doi: 10.1007/s00464-011-1639-8. Epub 2011 Apr 13. PMID 21487883
- [Background] Ford JA, Soop M, Du J, Loveday BP, Rodgers M. Systematic review of intraoperative cholangiography in cholecystectomy. Br J Surg. 2012 Feb;99(2):160-7. doi: 10.1002/bjs.7809. Epub 2011 Dec 19. PMID 22183717
- [Background] Agarwal BB. Patient safety in laparoscopic cholecystectomy. Arch Surg. 2009 Oct;144(10):979; author reply 979. doi: 10.1001/archsurg.2009.180. No abstract available. PMID 19841374
- [Background] Figueiredo JL, Siegel C, Nahrendorf M, Weissleder R. Intraoperative near-infrared fluorescent cholangiography (NIRFC) in mouse models of bile duct injury. World J Surg. 2010 Feb;34(2):336-43. doi: 10.1007/s00268-009-0332-8. PMID 20033407
- [Background] Figueiredo JL, Nahrendorf M, Vinegoni C, Weissleder R. Intraoperative near-infrared fluorescent cholangiography (NIRFC) in mouse models of bile duct injury: reply. World J Surg. 2011 Mar;35(3):694-5. doi: 10.1007/s00268-010-0728-5. No abstract available. PMID 20645091
- [Background] Tagaya N, Shimoda M, Kato M, Nakagawa A, Abe A, Iwasaki Y, Oishi H, Shirotani N, Kubota K. Intraoperative exploration of biliary anatomy using fluorescence imaging of indocyanine green in experimental and clinical cholecystectomies. J Hepatobiliary Pancreat Sci. 2010 Sep;17(5):595-600. doi: 10.1007/s00534-009-0195-2. Epub 2009 Oct 6. PMID 19806299
- [Background] Matsui A, Tanaka E, Choi HS, Winer JH, Kianzad V, Gioux S, Laurence RG, Frangioni JV. Real-time intra-operative near-infrared fluorescence identification of the extrahepatic bile ducts using clinically available contrast agents. Surgery. 2010 Jul;148(1):87-95. doi: 10.1016/j.surg.2009.12.004. Epub 2010 Feb 1. PMID 20117813
- [Background] Ishizawa T, Bandai Y, Ijichi M, Kaneko J, Hasegawa K, Kokudo N. Fluorescent cholangiography illuminating the biliary tree during laparoscopic cholecystectomy. Br J Surg. 2010 Sep;97(9):1369-77. doi: 10.1002/bjs.7125. PMID 20623766
- [Background] Ishizawa T, Kaneko J, Inoue Y, Takemura N, Seyama Y, Aoki T, Beck Y, Sugawara Y, Hasegawa K, Harada N, Ijichi M, Kusaka K, Shibasaki M, Bandai Y, Kokudo N. Application of fluorescent cholangiography to single-incision laparoscopic cholecystectomy. Surg Endosc. 2011 Aug;25(8):2631-6. doi: 10.1007/s00464-011-1616-2. Epub 2011 Mar 18. PMID 21424202
- [Background] Aoki T, Murakami M, Yasuda D, Shimizu Y, Kusano T, Matsuda K, Niiya T, Kato H, Murai N, Otsuka K, Kusano M, Kato T. Intraoperative fluorescent imaging using indocyanine green for liver mapping and cholangiography. J Hepatobiliary Pancreat Sci. 2010 Sep;17(5):590-4. doi: 10.1007/s00534-009-0197-0. Epub 2009 Oct 21. PMID 19844652
- [Background] Schols RM, Bouvy ND, Masclee AA, van Dam RM, Dejong CH, Stassen LP. Fluorescence cholangiography during laparoscopic cholecystectomy: a feasibility study on early biliary tract delineation. Surg Endosc. 2013 May;27(5):1530-6. doi: 10.1007/s00464-012-2635-3. Epub 2012 Oct 18. PMID 23076461
- [Background] Mitsuhashi N, Kimura F, Shimizu H, Imamaki M, Yoshidome H, Ohtsuka M, Kato A, Yoshitomi H, Nozawa S, Furukawa K, Takeuchi D, Takayashiki T, Suda K, Igarashi T, Miyazaki M. Usefulness of intraoperative fluorescence imaging to evaluate local anatomy in hepatobiliary surgery. J Hepatobiliary Pancreat Surg. 2008;15(5):508-14. doi: 10.1007/s00534-007-1307-5. Epub 2008 Oct 4. PMID 18836805
- [Background] Ashitate Y, Stockdale A, Choi HS, Laurence RG, Frangioni JV. Real-time simultaneous near-infrared fluorescence imaging of bile duct and arterial anatomy. J Surg Res. 2012 Jul;176(1):7-13. doi: 10.1016/j.jss.2011.06.027. Epub 2011 Jul 14. PMID 21816414
- [Background] Schols RM, Bouvy ND, van Dam RM, Masclee AA, Dejong CH, Stassen LP. Combined vascular and biliary fluorescence imaging in laparoscopic cholecystectomy. Surg Endosc. 2013 Dec;27(12):4511-7. doi: 10.1007/s00464-013-3100-7. Epub 2013 Jul 23. PMID 23877766
- [Derived] van den Bos J, Schols RM, Luyer MD, van Dam RM, Vahrmeijer AL, Meijerink WJ, Gobardhan PD, van Dam GM, Bouvy ND, Stassen LP. Near-infrared fluorescence cholangiography assisted laparoscopic cholecystectomy versus conventional laparoscopic cholecystectomy (FALCON trial): study protocol for a multicentre randomised controlled trial. BMJ Open. 2016 Aug 26;6(8):e011668. doi: 10.1136/bmjopen-2016-011668. PMID 27566635